CLINICAL TRIAL: NCT03421158
Title: Comparing the Analgesic Effects of Four Non-pharmacological Interventions on Term Newborns Undergoing Heel Lance
Brief Title: Non-pharmacological Analgesic Effects on Term Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Annette Nasr, Clinical Assistant Professor, Pediatrics, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31216
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2017-12

CONDITIONS: Pain; Breast Feeding
Keywords: neonates; Non-pharmacological
MeSH Terms: conditions — Pain; Breast Feeding | interventions — Lactation; Sucrose; Pacifiers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (No Intervention): Newborns received no pain interventions during the procedure
- Breastfeeding (Experimental): Newborns were breastfed during the procedure
  Interventions: Behavioral: breastfeeding
- Oral Sucrose (Experimental): Newborns were given oral sucrose during the procedure
  Interventions: Dietary Supplement: oral sucrose
- Skin to skin contact (Experimental): Newborns were placed in direct contact with their mothers during the procedure
  Interventions: Behavioral: Skin-to-Skin contact
- Non-nutritive sucking (Experimental): Newborns were given a pacifier to suck on during the procedure
  Interventions: Behavioral: Non-nutritive sucking

INTERVENTIONS:
Behavioral: breastfeeding — Newborns were breastfed during the procedure
  Arms: Breastfeeding
Dietary Supplement: oral sucrose — Newborns were given oral sucrose during the procedure
  Arms: Oral Sucrose
Behavioral: Skin-to-Skin contact — Newborns were placed in direct contact with their mothers during the procedure
  Arms: Skin to skin contact
Behavioral: Non-nutritive sucking — newborns were given a pacifier to suck on during the procedure
  Other Names: Pacifier
  Arms: Non-nutritive sucking

SUMMARY:
The purpose of this study is to compare the analgesic effects of four non-pharmacological interventions: skin-to-skin contact, breastfeeding, oral sucrose and nonnutritive sucking in newborns receiving a heel lance procedure.

DETAILED DESCRIPTION:
This is an randomized control clinical study. study population is healthy term newborns.Patients were identified by chart review and consent was received by nurse researcher. Newborns were randomized into either the control group who received no pain intervention or the intervention group who received one of four non-pharmacological pain interventions: skin to skin contact, breastfeeding, oral sucrose, and nonnutritive sucking.

A heel lance for newborn screen blood sampling was selected as a study procedure and performed by a hospital technician following standard protocol. Pain scoring was assessed by two research nurses after the hell lance and through the procedure. Neonatal Pain, Agitation and Sedation Scale (NPASS) was selected as a pain assessment tool for this study.

The average pain score from two research nurses were used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Gestational Age 38-40
* 2.5-4.0kg
* 24-48hours of age
* Receiving heel lance procedure
* Apgar>7 at birth
* NPASS<3 at time of heel lance

Exclusion Criteria:

* Prior heel lance procedure
* birth trauma
* forceps or vacuum delivery
* maternal drug abuse during delivery

Ages: 24 Hours to 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 236 (Actual)
Dates: Start 2014-11-07 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Decrease in Neonatal Pain, Agitation and Sedation Scale (NPASS) scores for newborns receiving non-pharmacologic interventions | 12 month
  Neonatal Pain, Agitation and Sedation Scale (NPASS) measures both behavioral and physiological components of pain by evaluating five key elements, and scores pain from 0-10 (Patricia A. Hummel, 2004). The assessment criteria are crying irritability, behavior state, facial expression, extremities tone, and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Chang, BSN,MD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: Yes